CLINICAL TRIAL: NCT03764917
Title: Study on the Effect of NGS Combined With RNAseq on Tumor Immune Escape in Advanced Non-small Cell Lung Cancer EGFR and ALK Mutant Negative Patients
Brief Title: NGS Combined With RNAseq on Tumor Immune Escape in NSCLC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Prof. Caicun Zhou, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: YS2018-003
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NGS; RNAseq
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Time — Different detecting time

SUMMARY:
Study on the tumor immune escape in advanced non-small cell lung cancer patients with EGFR and ALK mutant negative by NGS combined with RNAseq

DETAILED DESCRIPTION:
Study on the tumor immune escape in advanced non-small cell lung cancer patients with EGFR and ALK mutant negative by NGS combined with RNAseq. Detecting non-small cell lung cancer patient NGS and RNAseq data before first-line chemotherapy, after two cycles chemotherapy and after disease progression.

ELIGIBILITY:
Inclusion Criteria:

Non-small cell lung cancer patient First-line chemotherapy with platinum-based chemotherapy

Exclusion Criteria:

EGFR mutant positive Alk mutant positive

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patient First-line chemotherapy with platinum-based chemotherapy Without EGFR and Alk mutation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
numbers of immune cells | 24 months
  detecting numbers of immune cells before first-line chemotherapy, after two cycles chemotherapy and after disease progression

SECONDARY OUTCOMES:
numbers of tumor mutations | 24 months
  detecting numbers of tumor mutations before first-line chemotherapy, after two cycles chemotherapy and after disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Yayi He, MD, PHD, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He Y, Chen L, Zhao L, Dang S, Liu G, Sasada S, Ma PC, van Zandwijk N, Rosell R, Popper HH, Wang H, Jiang M, Guo H, Liu X, Chen S, Zhang X, Xu M, Zhu B, Liu M, Zhou C. Genomic and transcriptional alterations in first-line chemotherapy exert a potentially unfavorable influence on subsequent immunotherapy in NSCLC. Theranostics. 2021 May 13;11(14):7092-7109. doi: 10.7150/thno.58039. eCollection 2021. PMID 34093873